CLINICAL TRIAL: NCT00839306
Title: A Randomized Double-Blind Parallel Study of Rabeprazole Extended Release 50 mg Versus Ranitidine 150 mg for Maintenance of Healed Erosive Gastroesophageal Reflux Disease (GERD)
Brief Title: Rabeprazole Extended Release 50 mg Versus Ranitidine 150 mg for Maintenance of Healed Erosive Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-G000-306
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal; Reflux; Disease; GERD
MeSH Terms: conditions — Gastroesophageal Reflux; Disease | interventions — Rabeprazole; Ranitidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Rabeprazole ER
- 2 (Active Comparator)
  Interventions: Drug: Ranitidine

INTERVENTIONS:
Drug: Rabeprazole ER — 50 mg capsule, taken orally, once daily for 26 weeks.
  Other Names: Aciphex
  Arms: 1
Drug: Ranitidine — 150 mg capsule, taken orally, twice daily for 26 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy of rabeprazole extended release 50 mg (once daily) versus ranitidine 150 mg (twice daily) in the maintenance of complete healing in subjects with healed erosive gastroesophageal reflux disease (eGERD).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, double-dummy, parallel-group study. Subjects who meet all eligibility criteria will be randomly assigned to 1 of 2 treatment groups, rabeprazole extended release 50 mg (once daily) or ranitidine 150 mg (twice daily).

Please note that this study is not a duplicate of E3810-G000-305; this is a separate study being conducted along with -305.

ELIGIBILITY:
KEY INCLUSION CRITERIA:

1. Prior completion of Study E3810-G000-302 or -303. Subjects will need to have healed erosive esophagitis (absence of esophageal mucosal breaks or erosions) confirmed by EGD and sustained resolution of heartburn at Visit 4 or 5 of Study E3810-G000-302 or -303.

KEY EXCLUSION CRITERIA:

1. Esophageal motility disorders (achalasia, scleroderma, or esophageal spasm).
2. Barrett's esophagus or esophageal stricture.
3. Use of prescription or non-prescription proton pump inhibitors (PPIs), histamine receptor antagonists (H2RA), antacids, sucralfate, misoprostol, prokinetics or drugs with significant anticholinergic effects throughout the study.
4. Subjects who require chronic use of nonsteroidal anti-inflammatory drugs (NSAIDs), oral steroids (>= 20 mg/day prednisone or equivalent), or aspirin (->; 325 mg/day).
5. Significant hepatic, renal, respiratory, endocrine, hematologic, neurologic, psychiatric, or cardiovascular system abnormalities that would be likely to interfere with the conduct of the study, the interpretation of study results, or the health of the subject during the study.
6. Any condition that would make the subject, in the opinion of the Investigator or Sponsor, unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Rossiter, M.D., Study Director — Eisai Inc.
Locations (4):
- United States (4):
  - Associates, Ltd., Moline, Illinois
  - Midwest Clinical, Moline, Illinois
  - Research, Moline, Illinois
  - Moline, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible for this study if they had completed one of the healing studies (E3810-G000-302 or E3810-G000-303), had no evidence of oesophageal erosions, had sustained heartburn resolution, and had no record of any serious adverse event (SAE) related to study medication during the healing study.
Pre-assignment Details: Out of 240 participants who were randomized in this study, 237 participants received study treatment.
Groups:
- RAN 150mg BID: Morning dose included 1 x Placebo to match RAB (Rabeprazole) ER (Extended Release) 50mg capsule and 1 x RAN (Ranitidine) 150mg capsule. Evening dose included 1 x RAN 150mg capsule. Received study drug orally daily for 26 weeks.
- RAB ER 50mg QD: Morning dose included 1 x RAB ER 50mg capsule and 1 x Placebo to match RAN 150mg capsule. Evening dose included 1 x Placebo to match RAN 150mg capsule. Received study drug orally daily for 26 weeks.
Period: Overall Study
Arm/Group | RAN 150mg BID | RAB ER 50mg QD
Started | 60 (Treated) | 177 (Treated)
Completed | 35 | 134
Not Completed | 25 | 43
Not completed — Adverse Event | 3 | 5
Not completed — Lost to Follow-up | 6 | 9
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Lack of Efficacy | 5 | 4
Not completed — Other | 6 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RAN 150mg BID | RAB ER 50mg QD | Total
Number analyzed (Participants) | 60 | 177 | 237
Age, Customized [Mean (Standard Deviation); unit: Years] | 47.5 (13.55) | 47.5 (12.06) | 47.5 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 88 | 116
  Male | 32 | 89 | 121

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Investigator-recorded Sustained Resolution of Heartburn at Week 26
Description: Heartburn or other GERD-associated symptoms (regurgitation, epigastric or chest pain, dysphagia, belching, bloating, early satiety, other) was based on a 4-point Likert scale that included the following: None (No symptoms); Mild (Awareness of symptoms but easily tolerated); Moderate (Discomforting symptom sufficient to cause interference with normal activities including sleep); Severe (Incapacitating symptom, inability to perform normal activities).
Time Frame: Baseline to Week 26
Population: ITT
Measure: Number; unit: Percentage of Participants
Groups:
- RAB ER 50mg QD: Morning dose included 1 x RAB ER 50mg capsule and 1 x Placebo to match RAN 150mg capsule. Evening dose inlcuded 1 x Placebo to match RAN 150mg capsule. Received study drug orally daily for 26 weeks.
Arm/Group | RAN 150mg BID | RAB ER 50mg QD
Number analyzed (Participants) | 60 | 177
Percentage of Participants
  Yes | 8.3 | 53.7
  No | 16.7 | 17.5
  Missing | 75 | 28.8

2. Primary Outcome: Percentage of Participants With Maintenance of Complete Healing of eGERD at Week 26
Description: eGERD (erosive gastroesophageal reflux disease) healing measured by the Time-to-Relapse of Oesophageal Erosions using an Esophagogastroduodenoscopy (EGD). Lesions were identified and graded using the following Los Angeles (LA) classification of Oesophagitis: Not Present: No breaks (erosions) in the oesophageal mucosa (however, edema, erythema, or friability may be present).
  Grade A: One or more mucosal breaks not more than 5mm in maximum length. Grade B: One or more mucosal breaks more than 5mm in maximum length, but not continuous between the tops of 2 mucosal folds.
  Grade C: Mucosal breaks continuous between the tops of 2 or more mucosal folds, but involving less than 75% of the esophageal circumference.
  Grade D: Mucosal breaks involving at least 75% of the esophageal circumference.
Time Frame: Baseline to Week 26
Population: Intent-to-Treat (ITT) Population - all randomized subjects who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | RAN 150mg BID | RAB ER 50mg QD
Number analyzed (Participants) | 60 | 177
Percentage of Participants | 31.7 | 88.4

ADVERSE EVENTS:
Time Frame: For each participant, from the time of administration of the first dose of study drug up to 30 days after the administration of the last dose of study drug or up to resolution of adverse event or up to approximately 30 weeks.
Description: Data are presented as number of participants with treatment emergent adverse events (serious and nonserious). The analysis was performed using the Safety Analysis Set (SAS), defined as all subjects who received at least 1 dose of study drug and had a postbaseline safety assessment.
Arm/Group | RAN 150mg BID | RAB ER 50mg QD
Serious Adverse Events (participants affected / at risk) | 1/56 | 3/170
Other Adverse Events (participants affected / at risk) | 22/56 | 42/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAN 150mg BID (N=56) | RAB ER 50mg QD (N=170)
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAN 150mg BID (N=56) | RAB ER 50mg QD (N=170)
Gastritis (Gastrointestinal disorders) | 4 | 17
Sinusitis (Infections and infestations) | 1 | 10
Hiatus hernia (Gastrointestinal disorders) | 6 | 7
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Erosive oesophagitis (Gastrointestinal disorders) | 5 | 2
Acquired oesophageal web (Gastrointestinal disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No